CLINICAL TRIAL: NCT01893788
Title: Eplerenone and Aliskiren Research Targeting Hypertensive Patients With Left Ventricular Hypertrophy
Acronym: EARTH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nagoya University (Other)
Responsible Party: Principal Investigator, TOYOAKI MUROHARA, Professor of Medicine, Nagoya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nagoya University
Record Dates: First submitted 2013-04-30; First posted 2013-07-09 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Hypertensive Left Ventricular Hypertrophy
Keywords: hypertension; left ventricular hypertrophy; renin angiotensin system; aldosterone; aliskiren; eplerenone; P3NP
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — aliskiren; Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Active Comparator): Aliskiren group treated with 150-300mg daily aliskiren without diuretics or ACE inhibitors or angiotensin receptor blockers.
  Interventions: Drug: Aliskiren
- Eplerenone (Active Comparator): Eplerenone group treated with 50-100mg daily eplerenone without diuretics or ACE inhibitors or angiotensin receptor blockers
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Aliskiren — Aliskiren: 150 to 300 mg daily for 48 weeks
  Other Names: Rasilez
  Arms: Aliskiren
Drug: Eplerenone — 50 to 100 mg daily for 48 weeks
  Other Names: Selara
  Arms: Eplerenone

SUMMARY:
The primary objective of this study is to determine which treatment will be more effective to reduce left ventricular mass in hypertensive patients with left ventricular hypertrophy comparing aliskiren and eplerenone.

ELIGIBILITY:
Inclusion Criteria:

Male or female ≧ 20 years of age Clinical diagnosis of hypertension Patients who are able to provide written informed consent

Exclusion Criteria:

1. History of congestive heart failure, myocardial infarction, or coronary revascularization in the recent 6 months.
2. Planned to taking percutaneous coronary intervention and coronary artery bypass graft
3. Severe hypertension (≧ 180/110 mmHg) or secondary hypertension or malignant hypertension.
4. History of stroke, cerebral hemorrhage, subarachnoid hemorrhage, transient ischemic attack in the recent 6 months
5. Severe valvular heart disease or atrial fibrillation
6. Congenital heart disease
7. Severe heart failure (NYHA functional class Ⅳ)
8. Current treatment with aliskiren or eplerenone or diuretics
9. Taking potassium preparation or potassium-sparing diuretic
10. Estimated GFR ≦ 30ml/min/1.73m２ at screening or current treatment with hemodialysis
11. Potassium > 5.0mEq/L at screening
12. Diabetes mellitus with microalbuminuria or albuminuria
13. Impairment of liver function (liver failure, liver cirrhosis)
14. Pregnant woman or possibly pregnant woman
15. History of malignant tumor include hematological neoplasm
16. Current treatment with itraconazole, cyclosporin, ritonavir or nelfinavir
17. Prior treatment with, hypersensitivity to, intolerance of or contra-indication to aliskiren and/or eplerenone
18. Current participation in another clinical trial
19. Serious non-cardiovascular disease severely limiting life expectancy
20. Contra-indication to MRI

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
reduction of left ventricular hypertrophy measured by magnetic resonance imaging | 12 month
  To compare the 12 month left ventricular mass or left ventricular mass and index measured by magnetic resonance imaging with baseline.

SECONDARY OUTCOMES:
Cardiovascular events | 12 month
  total death, composite cardiovascular events, cardiac function eveluated by UCG,reduction of left ventricular hypertrophy measured by UCG

OTHER OUTCOMES:
Biochemical parameters | 12 month
  BNP, PIIINP etc

CONTACTS AND LOCATIONS:
Overall Officials: Toyoaki Murohara, MD, PhD, Principal Investigator — Department of Cardiology, Nagoya University Graduate School of Medicine
Locations (1):
- Department of Cardiology, Nagoya University Graduate School of Medicine, Nagoya, Aichi-ken, Japan